CLINICAL TRIAL: NCT03950414
Title: A Phase I Dose-Escalation Study Evaluating Safety and Tolerability of Viral-Specific T Cells Against CMV in Adult Solid Organ Transplant Recipients
Brief Title: A Dose-Escalation Study Evaluating Safety and Tolerability of Viral-Specific T Cells Against CMV in Adult Solid Organ Transplant Recipients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Patient Population
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0060; PACT VST-C-002 (Other Grant/Funding Number: GALIPEAU SMPH START UP-PACT SUPPORT); Protocol Version 11/1/2021 (Other: UW Madison)
Record Dates: First submitted 2019-04-15; First posted 2019-05-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cytomegalovirus Infections; Solid Organ Transplant
Keywords: T-cell; immunotherapy
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: 3+3 dose-escalation, open label, non-randomized, non-placebo controlled, single group assignment study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tier 1 (Experimental): 3 participants enrolled at dose level 5x10^3 cells/kg of CMV viral specific T-cells
  Interventions: Biological: CMV specific T-cells

INTERVENTIONS:
Biological: CMV specific T-cells — Naturally occurring, allogeneic donor lymphocytes derived from a leukapheresis or a whole blood product, enriched for CMV-specific CD4+ and CD8+ T cells Suspension of CMV-specific T cells in 10 mL of 0.9% NaCl with 2% Human Serum Albumin(HSA) via IV bolus injection
  * Low Dose Tier - Viral-Specific T cell infusion 5 x10^3 cells/kg body weight(BW)
  * Mid Dose Tier - Viral-Specific T cell infusion 1.25 x10^4 cells/kg BW
  * High Dose Tier - Viral-Specific T cell infusion 2.5 x10^4 cells/kg BW Product will be administered fresh intravenously to recipient within four hours of collection.

SUMMARY:
This study measures the tolerability of viral-specific T cells against Cytomegalovirus (CMV) in adult solid organ transplant (SOT) recipients. Participants are expected to be on study for 52 +/- 3 weeks.

DETAILED DESCRIPTION:
Viral infections, or their reactivation in the immunocompromised host, remain serious complications that adversely affect outcomes of transplantation. These infections may be refractory to pharmacologic treatment and result in increased morbidity and mortality after transplantation. Furthermore, the available pharmacologic therapies can result in severe toxicities.

Once an infection occurs, adequate immune reconstitution is decisive for recovery from viral disease after solid organ transplantation. The present trial will consist of the treatment of solid organ transplant recipients diagnosed with severe CMV infection when standard antiviral therapy is ineffective (disease progression on therapy, decline in viral load less than 10-fold in 2 weeks, known drug resistance), or toxic (end-organ damage), with virus-specific T cells using the CliniMACS® Prodigy System. These are the patients with the greatest unmet need and greatest risk or morbidity and allograft loss due to CMV infection. CMV-specific T cells will be isolated from donor leukapheresis products using the CliniMACS® Prodigy. Prior studies on transfer of CMV-specific T cells have been shown to be safe and efficacious in the treatment of CMV infections.

The primary objective of this Phase I trial is to evaluate the safety and tolerability of CMV-specific T-cell transfer in adult patients suffering from CMV infections following solid organ transplantation using a dose escalation design. The incubation with viral antigens (MACS GMP PepTivator) allows the enrichment of CMV-specific CD4+(Cluster of Differentiation 4) and CD8+(Cluster of Differentiation 8) T cells. Increasing evidence of the safety and efficacy of CMV-specific T-cell is available. Furthermore, the safety and efficacy of the specific manufacturing approach using the fully automated protocol of the ClinMACS® Prodigy for the isolation of CMV-specific T cells against CMV has been described and demonstrated that these cells retain their biological properties.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18 and ≤75) patients suffering from CMV reactivation/infections following solid organ transplantation (e.g., liver, pancreas, lung, heart, and multi-solid organ)

   * CMV reactivation/viremia defined as positive (>250 copies/mL) CMV qPCR(quantitative polymerase chain reaction) AND/OR
   * Presence of symptoms secondary to CMV infection or evidence of invasive CMV infection (e.g. pneumonitis, colitis)

   AND ONE OF THE FOLLOWING CRITERIA:
   * Absence of an improvement of viral load after ≥ 14 days of standard antiviral therapy with ganciclovir, valganciclovir or foscarnet (decrease by at least 1 log, i.e. 10-fold), or
   * New, persistent and/or worsening CMV-related symptoms, signs and/or markers of end organ compromise while on anti-viral therapy with medications such as ganciclovir, acyclovir, valganciclovir, foscarnet, cidofovir, IVIG(Intravenous immunoglobulin), and/or letermovir, or
   * Have contraindications or experience adverse effects of anti-viral therapy with medications such as ganciclovir, acyclovir, valganciclovir, foscarnet, cidofovir, IVIG, and/or letermovir, or
   * Known resistance to the anti-viral medications ganciclovir, foscarnet and/or cidofovir based on molecular testing
2. Availability of eligible donor
3. Written informed consent given by patient

Exclusion Criteria:

1. Patient with acute rejection of allograft at time of T-cell transfer
2. Patient receiving steroids (>0.5 mg/kg body weight (BW) prednisone equivalent) at the time of T-cell transfer
3. Patient treated with Thymoglobulin (ATG), Alemtuzumab or T-cell immunosuppressive monoclonal antibodies within 28 days
4. Patients with CMV retinitis
5. Concomitant enrollment in another clinical trial interfering with endpoints of this study
6. Any medical condition which could compromise participation in the study according to the investigator's assessment
7. Known HIV infection
8. Female patient who is pregnant or breast-feeding, or adult of reproductive potential not willing to use an effective method of birth control during study treatment Note: Women of childbearing potential must have a negative serum pregnancy test at study entry.
9. Patients unwilling or unable to comply with the protocol or unable to give informed consent

Donor Eligibility

Donor selection priority: The original donor will be the first choice as the source of T cells. If donation from the original organ donor is not possible (e.g., donor is unavailable or ineligible), then an alternative related donor will be selected, with preference for those who have full HLA matching in 6/6 loci over those with partial HLA matching (≥ 2/6 HLA loci). See Appendix 1 for patient and donor screening procedures.

1. ≥ 18 years old
2. Available and capable of undergoing a single standard 2 blood volume leukapheresis or donation of one unit of whole blood.
3. If the original transplant donor is not eligible, then an eligible fully matched or eligible partially matched family member will be used as the donor.
4. Related donors must be at least partially HLA compatible, matching with recipient in at least 2/6 HLA loci (HLA-A, HLA-B and HLA-DRB1 will be considered for this).
5. Donors must be CMV IgG seropositive.
6. Donors must show CMV T-cell activation after incubation with MACS GMP PepTivator Peptide Pools of CMV pp65 before undergoing leukapheresis.
7. Donor must meet the criteria for donor selection defined in the UWHC Hematopoietic Stem Cell Transplant Program SOP and FACT standards, which comply with 21 CFR 1271, subpart C.
8. Donor must provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability:Time of Occurence of Acute GVHD | up to 15 weeks
  Time to occurrence of acute GVHD of any grade will be evaluated using the Kaplan-Meier method to assess incidence and severity of acute GVHD from day of T-cell transfer. The first day of GVHD onset at a certain grade will be used to calculate a cumulative incidence curve for that GVHD grade. Overall, cumulative incidence curves will be computed along with the 95% confidence intervals until Week 12 after T-cell transfer with death considered as a competing risk.
Safety and Tolerability: Number of infusion-related adverse events | up to 7 weeks
  Incidence of grades 3-5 infusion-related adverse events, grades 4-5 non-hematological adverse events within four weeks of the CMV-VST dose that are not due to the pre-existing infection or original malignancy or pre-existing co-morbidities
Incidence of acute infusion-related toxicity | from T-cell transfer to 4 hours post injection, upto 3 weeks
  Incidence of acute infusion-related toxicity as assessed by maximum toxicity on the day of T-cell transfer, evaluated by measuring vital signs prior to and at different times after the T-cell transfer and monitoring of specific adverse events (chills, nausea, vomiting, diarrhea, abdominal pain, allergic reactions, respiratory dysfunction or headache from T-cell transfer to 4 hours post injection)
Severity of acute infusion-related toxicity as measured by Cytokine release syndrome (CRS) Grading criteria | from T-cell transfer to 4 hours post injection, upto 3 weeks
  Severity of acute infusion-related toxicity will be assessed by CRS grading criteria.
  Grade 1 Symptoms are not life threatening and require symptomatic treatment only, (e.g., fever, nausea, fatigue, headache, myalgias, malaise) Grade 2 Symptoms require and respond to moderate intervention Grade 3 Symptoms require and respond to aggressive intervention Grade 4 Life-threatening symptoms Grade 5 Death
  Any grade 3 or greater occurrence of CRS will be considered a serious adverse event for this study.
Number of Participants of Newly Occurring Acute Rejection after T-cell Transfer | up to 15 weeks
  Incidence and severity of acute rejection of the organ allograft will in part be measured by number of participants of newly occurring acute rejection after T-cell transfer
Incidence of de novo Antibodies against Organ Allograft Donor (dnDSA) after T-cell Transfer | up to 55 weeks
  Incidence and severity of acute rejection of the organ allograft will in part be measured by presence of de novo antibodies against organ allograft donor (dnDSA) after T-cell transfer
Incidence of GVHD Grade ≥1 | up to 15 weeks
  Incidence and severity of Graft-versus-host disease (GVHD) will be measured by occurrence of acute GVHD grade ≥1 or aggravation of pre-existing acute GVHD after T-cell transfer

SECONDARY OUTCOMES:
Feasibility: Was production of CMV Virus specific T lymphocyte (VST) from donors accomplished? | up to 3 weeks
  There is no minimum cell count required for the study as it can vary. Successful production of CMV Virus specific T lymphocyte (VST) from donors will be tracked by a Yes/No question.
  Production of cell accomplished: yes/no
Feasibility: Participant Drop-out rate | up to 3 weeks
  Evaluation of feasibility of CMV specific T cell transfer in adult patients suffering from severe CMV infection following solid organ transplantation in part will be measured by participant drop out rate
Feasibility: Time from patient inclusion to administration of CMV-VST | up to 21 days
  Evaluation of feasibility of CMV specific T cell transfer in adult patients suffering from severe CMV infection following solid organ transplantation in part will be measured by the amount of time from patient inclusion to administration of CMV-VST
Efficacy: Percentage of patients with ≥1 log decrease in CMV viral load | up to 15 weeks
  Evaluation of efficacy of CMV-specific T-cell transfer in adult patients suffering from severe CMV infection following solid organ transplantation in part will be measured in terms of percentage of patients with ≥1 log decrease in CMV viral load at Week 12
Efficacy:Time to 1 log change in CMV viral load | up to 15 weeks
  Evaluation of efficacy of CMV-specific T-cell transfer in adult patients suffering from severe CMV infection following solid organ transplantation in part will be measured in terms of time to 1 log change in CMV viral load
Efficacy:Number of Participants with CMV clearance | up to 15 weeks
  Efficacy evaluation in part will be measured by number of participants with CMV clearance. Either negative polymerase chain reaction (PCR) or <250 copies/mL will be considered as CMV clearance.
Efficacy: Time of clearance of CMV | up to 55 weeks
  Efficacy evaluation in part will be measured by number of days to achieve CMV clearance. Either negative polymerase chain reaction [PCR] or <250 copies/mL)will be considered as CMV clearance.
Efficacy: Number of participants having CMV reactivation | up to 55 weeks
  Efficacy in part will be measured by number of participants with CMV reactivations following initial viral clearance
Efficacy: Overall Survival of Participant | up to 55 weeks
  Overall survival rate of participants will be measured by time from T-cell transfer to death, graft loss, or last follow-up throughout the study
Efficacy:Number of Participants with Clinical response/resolution of symptoms of underlying viral infection | up to 15 weeks
  Efficacy in part will be measured by number of patients with resolution of clinical symptoms of underlying CMV infection from Day 7 (Week 1) to Week 12 after T-cell transfer as compared to Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh Parajuli, MBBS, Principal Investigator — University of Wisconsin, Madison; Jacques Galipeau, MD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No